CLINICAL TRIAL: NCT00892385
Title: A Phase I Study of Methoxyamine and Temozolomide in Patients With Advanced Solid Tumors
Brief Title: Methoxyamine and Temozolomide in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE1Y05; P30CA043703 (NIH); CASE1Y05 (Other: Case Comprehensive Cancer Center); WIRB-20070151 (Other: Western Institutional Review Board); NCI-2009-01286 (Registry Identifier: NCI)
Record Dates: First submitted 2009-05-01; First posted 2009-05-04 (Estimated); Last update posted 2019-02-22 (Actual); Status verified 2019-02

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — methoxyamine; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Non-CNS Disease (Experimental): A traditional 3 + 3 dose escalation design will be implemented. Successive cohorts of participants (3 participants/cohort) will be entered sequentially to each dose level. If 0/3 participants at a dose level experience dose limiting toxicity (DLT) new participants may be entered at the next higher dose level. If 1 participant has a DLT, 3 more will be enrolled at the same dose level. If the 1st participant in the expanded cohort (4th at the given DL), experiences no DLT, the remaining 2 participants can start treatment. If 2 or more experience DLT in the first cycle, no further participants are started at that dose and the MTD is the highest dose level in which <2 (of 6) participants develop DLT. If the final dose level is deemed the MTD, 6 participants will be treated at this dose level even if a DLT has not been observed.
  Interventions: Drug: Methoxyamine; Drug: Temozolomide
- CNS Disease (Experimental): A traditional 3 + 3 dose escalation design with successive cohorts of 3 participants will be entered sequentially to each dose level. If 0/3 participants experience DLT, new participants may be entered at the next higher dose level. If 1 participant has a DLT, 3 more will be enrolled at the same dose level. If the 1st participant in the expanded cohort (4th at the given DL), experiences no DLT, the remaining 2 participants can start treatment. If 1/3 participants experience a non-CNS DLT in Cohort B dose level 6, dose escalation will continue to dose level 7, as 3 subjects have already been treated in Cohort A dose level 6 and 7 subjects in Cohort A dose level 7, none of whom experienced non-CNS toxicities. If 2 or more experience DLT in cycle 1, no more participants are started at that dose and the MTD is the highest dose where <2/6 participants develop DLT. If the final dose level is deemed the MTD, 6 participants will be treated at this dose level even if no DLT has been observed.
  Interventions: Drug: Methoxyamine; Drug: Temozolomide

INTERVENTIONS:
Drug: Methoxyamine — For all cycles, TMZ will be given orally for 5 days every 28 days. MX will be given as a single one-hour IV infusion every 28 days. Temozolomide will be administered within 5 minutes following the initiation of methoxyamine.
  Other Names: NSC-3801; MX
Drug: Temozolomide — Patients receive oral temozolomide once daily on days 1-5. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Other Names: TMZ

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as methoxyamine and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving methoxyamine together with temozolomide may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of methoxyamine when given together with temozolomide in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the maximum tolerated dose of methoxyamine given in conjunction with temozolomide in patients with and without CNS disease.
* To determine the dose limiting toxicities of the combination of methoxyamine and temozolomide in patients with and without CNS disease.
* To determine the pharmacokinetics of these two agents when given alone or in combination, as well as the pharmacokinetic profile of methoxyamine after single one-hour IV administration.
* To determine relative DNA damage, as single or double strand breaks by comet assay in blood mononuclear cells which will serve as a surrogate for tumor response to the drug combination.

OUTLINE: This is a dose escalation study of methoxyamine.

Patients receive oral temozolomide for 5 days every 28 days and methoxyamine IV over 1 hour every 28 days. Methoxyamine IV administration will follow, within 5 minutes, initial administration of TMZ on day 1. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Blood samples are collected periodically for correlative studies. Samples are analyzed for methoxyamine and temozolomide pharmacokinetics, apurinic/apyrimidinic sites, and DNA strand break determination by comet assay.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a histologically confirmed solid tumor that is considered incurable and is not amenable to conventional surgical, radiation therapy or chemotherapy treatment programs.
* Prior chemotherapy and/or radiation are allowed. At least 3 weeks must have elapsed since prior large-field radiation therapy; patients must have been off previous anti-cancer therapy for at least 3 weeks (6 weeks for mitomycin-C and nitrosoureas); and recovered from all treatment related toxicity to < grade 1 according to NCI CTCAE version 3.0 (with the exception of alopecia and radiation-induced taste changes). Prior temozolomide treatment is not restricted.
* ECOG performance status (PS) 0-2 (Karnofsky PS 50-100%)
* Life expectancy ≥ 12 weeks
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count ≥ 1,500/μL
  * Platelet count ≥ 100,000/μL
  * Hemoglobin ≥ 10.0 g/dL
  * Total bilirubin ≤ 1.5 mg/dL
  * AST ≤ 2.5 times upper limit of normal
  * Creatinine ≤ 1.5 mg/dL and/or creatinine clearance ≥ 60 mL/min
* Patients with known primary or metastatic CNS disease, are eligible for participation in cohort B, but not in cohort A.
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients may not be receiving any other investigational agents or have received other investigational agents for at least 3 weeks.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant and lactating women are excluded from this study because the methoxyamine and temozolomide combination is likely to be teratogenic.
* NYHA classification III or IV heart disease
* Patients with known primary or metastatic CNS disease (cohort B) are not eligible if they have a mini mental status exam score < 15 or evidence of leptomeningeal disease.
* Patients with pre-existing neurologic toxicity > grade1 (as per CTCAE, version 3.0) are not eligible for participation in cohort A.
* Patients screened for participation in cohort B with pre-existing neurologic toxicity > grade 2 (as per CTCAE, version 3.0) are not eligible, unless pre-existing neurologic toxicity is documented in detail and patient's participation in the trial has been approved by the neuro-oncology team at participating institutions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-08-16 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-08 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of methoxyamine | Courses repeat every 28 days in the absence of unacceptable toxicity.
  A total of 38 patients were analyzed to determine the maximum tolerated dose of methoxyamine in this study and this was determined in the non-CNS arm. An initial 6 patients received treatment with continuous dosing of methoxyamine and based on an assessment of pharmacokinetics, in this group, the study was revised to administer methoxyamine as a bolus dose. Thirty-eight patients received this type of dosing.
Dose limiting toxicities of the combination of methoxyamine and temozolomide | Courses repeat every 28 days in the absence of unacceptable toxicity.
  The 38 patients receiving bolus dosing of methoxyamine in this trial were used to determine any dose limiting toxicities.
Pharmacokinetics methoxyamine and temozolomide, when given alone or in combination | Blood sampling during cycles 1 and 2 depending upon the PK data from initial subjects.
  Thirty-eight patients were analyzed per the schedule above (after an initial 6 patients treated per an alternative dosing schedule).

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Eads, MD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-18): https://cdn.clinicaltrials.gov/large-docs/85/NCT00892385/Prot_SAP_000.pdf